CLINICAL TRIAL: NCT03901768
Title: Effects of Combined Topical and Systemic Steroid Administrations on Better Early Postoperative Pain Management in Total Knee Arthroplasty: a Prospective Double-blinded Placebo Controlled Randomised Clinical Trial
Brief Title: Effects of Combined Topical and Systemic Steroid Administrations on Better Early Postoperative Pain Management in Total Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chan Ping-Keung, Honorary Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 18-234
Record Dates: First submitted 2019-03-29; First posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Total Knee Replacement
MeSH Terms: interventions — Dexamethasone; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group dexamethasone (Experimental): A syringe having 4ml of 4mg/ml of dexamethasone is used for intravenous injection
  Interventions: Drug: Dexamethasone
- Group triamcinolone (Experimental): 1ml of 40mg triamcinolone is mixed in the syringes containing solution for intrarticualar local infiltration. The solution is injected intraarticularly.
  Interventions: Drug: Triamcinolone
- Group dexamethasone with triamcinolone (Experimental): A syringe having 4ml of 4mg/ml of dexamethasone is used for intravenous injection. 1ml of 40mg triamcinolone is mixed in the syringes containing solution for intrarticualar local infiltration. The solution is injected intraarticularly.
  Interventions: Drug: Dexamethasone; Drug: Triamcinolone
- Placebo group (Placebo Comparator): A syringe having 4ml of saline is used for intravenous injection. 1ml of saline is mixed in the syringes containing solution for intrarticualar local infiltration. The solution is injected intraarticularly.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Dexamethasone — a syringe having 4ml of 4mg/ml of dexamethasone is used for intravenous injection.
  Arms: Group dexamethasone; Group dexamethasone with triamcinolone
Drug: Triamcinolone — 1ml of 40mg triamcinolone is mixed in the syringes containing solution for intrarticualar local infiltration. The solution is injected intraarticularly.
  Arms: Group dexamethasone with triamcinolone; Group triamcinolone
Drug: Placebos — A syringe having 4ml of saline is used for intravenous injection. 1ml of saline is mixed in the syringes containing solution for intrarticualar local infiltration. The solution is injected intraarticularly.
  Arms: Placebo group

SUMMARY:
With the aging of population, osteoarthritis of knees and hips has become major orthopaedic problems in Hong Kong. Osteoarthritis of knees and hips is associated with significant pain problems and functional disability. Total joint replacement is the ultimate surgical procedure to deal with such problems.

However total joint replacement is associated with significant tissue damage and post-operative pain problems, which would affect post-operative recovery and rehabilitation.

The primary aims of total knee replacement are improvement in functional activities and reducing pain due to degenerated knee joints. However, there are around 20-30% of patients would develop significant pain problems despite uncomplicated total knee replacement. It accounts for major post-operative problems and burdens.

Procedure specific analgesic method with multi-model analgesia technique is well-known to be useful in post-operative pain management, which reduces the post-operative pain score. Despite the use of multi-modal analgesic technique, pain after total joint replacement is still an unsolved issue. It prolongs the recovery period and increases post-operative analgesic consumption.

Dexamethasone is a glucocorticoid which is associated with anti-inflammatory response. It is well known to have prophylaxis effect on post-operative nausea and vomiting. Perioperative single dose of systemic dexamethasone have shown to be useful for reduction in pain and cumulative opioid consumption. Meta-analysis from De Oliveira et al supports that dexamethasone (up to 0.2 mg/kg) is a safe and effective multimodal pain strategy after surgical procedures. However, this dose recommendation is not surgery specific. Recently, one review also supports even higher systemic steroid dose to ameliorate post-operative pain after hip and knee surgery. This is based on 3 RCTs using high dose steroid (125 mg methylpresnisolone and 40mg dexamethasone). However, large-scale safety and dose-finding studies are warranted before final recommendations. In view of these, it is essential to have more RCTs evaluating the optimal dose of steroid for pain management after hip and knee surgery.

Chronic steroid use is known to be associated with infection and gastrointestinal bleeding. It is essential to evaluate the safety profile associated with the use of high dose steroid -- risk of infection, gastrointestinal bleeding and hyperglycaemia etc. Published reviews have not raised concerns with perioperative single-dose administration in surgical patients. For hyperglycemia, P. Hans et al have shown that after the use of 10 mg dexamethasone, blood glucose level was increased in non-diabetic and type 2 diabetic patients undergoing abdominal surgery, in which glucose level and percentage change of glucose level were significant higher in diabetic group with glucose level peaked at around 2 hours after injection. Recent study by Basem B. Abdelmalak et al have shown that there was a comparable dexamethasone-induced hyperglycemic response in the diabetic and non-diabetic groups. Nevertheless, there was dexamethasone-induced hyperglycaemia in both groups. Close monitoring of blood glucose and correction of hyperglycaemia in those patients are recommended.

In previous studies, high-dose dexamethasone has shown to be effective and safe to be administered. The addition of dexamethasone to the multi-model analgesia is associated with anti-inflammatory response, thus extending the analgesic effect period for up to 72 hrs as purposed to 24-48 hrs. However, the recommended dose of dexamethasone is not surgery-specific and needs more studies to define the optimal dose. Therefore, it is essential to have more RCTs which evaluate the optimal dose of steroid for better pain management after hip and knee surgeries.

Investigators have recently performed a study evaluating the effect of high-dose dexemathasone. It is shown that dexamethasone 16mg is effective in managing acute postoperative pain after total knee arthroplasty. Another study have been performed by investigators to show the effectiveness of local application of triamcinolone to surgical sites after total knee arthroplasty.

In view of the above findings, the aim of this study is to compare the effect of intravenous dexamethasone, local application of triamcinolone and combined use of intravenous dexamethasone and local application of triamcinolone after total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Age 18-80 years old (For patients recruited from the Duchess of Kent Children's Hospital at Sandy Bay, they will also be aged from 18 to 80 years old)
* Scheduled for elective primary unilateral total knee replacement
* Chinese patients
* Able to speak and understand Cantonese
* Able to provide informed oral and written consent

Exclusion Criteria:

* Revision total knee replacement
* Single stage bilateral total knee replacement
* Known allergy to opioids, local anaesthetic drugs, paracetamol, non-steroidal anti-inflammatory drugs (NSAIDS) including COX-2 inhibitors
* History of chronic pain other than chronic knee pain
* History of insulin dependent diabetic mellitus, but not diabetic mellitus on oral hyperglycaemic agents
* History of hepatitis B or C carrier
* History of peptic ulcer
* Hx of tuberculosis
* History of immunosuppression
* Daily use of glucocorticoids
* Daily use of strong opioids (morphine, fentanyl, hydromorphone, ketobemidone, methadone, nicomorphine, oxycodone, or meperidine)
* History of severe heart disease (NYHA 2)
* Alcohol or drug abuse
* Impaired renal function, defined as preoperative serum creatinine level over 120 micromol/L
* Pre-existing neurological or muscular disorders
* Psychiatric illness or neurologic or psychiatric diseases potentially influencing pain perception
* Impaired or retarded mental state
* Difficulties in using patient controlled analgesia (PCA)
* Pregnancy
* Local infection
* On immunosuppresants
* Patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-04-26 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Pain (rest, moment) | From day 0 to 12 months after surgery
  Numeric rating scale is used to assess pain intensity in persons who are able to self report. It ranges from 0 to 10. Pain increases with the number.
PCA morphine consumption | From day 0 to the day on which patient was discharged from the hospital, assessed up to day 7
  Number of demands and goods
Active and passive ROM of knee (flexion and extension) | From day 0 to 12 months after surgery
  Active and passive range of motion of knee (flexion and extension)
Local Knee function e.g. KSKS | From day 0 to 12 months after surgery
  Knee society knee score is a total score which rates the knee joint and its function. Higher score represents better knee recovery. It ranges from 0 to 100. Total score is the sum of subscores. Subscales are pain, passive range of motion, stabilty, fixed flexion contracture, extension lag and alignment. Pain ranges from 0 to 50. Higher score represents milder pain. Passive range of motion ranges from 0 to 25. Higher score represents better recovery. Stability ranges from 0 to 25. Higher score represents better recovery. Fixed flexion contracture ranges from 0 to -15. Lower score represents worse recovery. Extension lag ranges from 0 to -15. Lower score represents worse recovery. Alignment ranges from 0 to -20. Lower score represents worse recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopaedics and Traumatology, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Oliveira GS Jr, Almeida MD, Benzon HT, McCarthy RJ. Perioperative single dose systemic dexamethasone for postoperative pain: a meta-analysis of randomized controlled trials. Anesthesiology. 2011 Sep;115(3):575-88. doi: 10.1097/ALN.0b013e31822a24c2. PMID 21799397
- [Background] Waldron NH, Jones CA, Gan TJ, Allen TK, Habib AS. Impact of perioperative dexamethasone on postoperative analgesia and side-effects: systematic review and meta-analysis. Br J Anaesth. 2013 Feb;110(2):191-200. doi: 10.1093/bja/aes431. Epub 2012 Dec 5. PMID 23220857
- [Background] Lunn TH, Kehlet H. Perioperative glucocorticoids in hip and knee surgery - benefit vs. harm? A review of randomized clinical trials. Acta Anaesthesiol Scand. 2013 Aug;57(7):823-34. doi: 10.1111/aas.12115. Epub 2013 Apr 15. PMID 23581549
- [Background] Srinivasa S, Kahokehr AA, Yu TC, Hill AG. Preoperative glucocorticoid use in major abdominal surgery: systematic review and meta-analysis of randomized trials. Ann Surg. 2011 Aug;254(2):183-91. doi: 10.1097/SLA.0b013e3182261118. PMID 21694581
- [Background] Salerno A, Hermann R. Efficacy and safety of steroid use for postoperative pain relief. Update and review of the medical literature. J Bone Joint Surg Am. 2006 Jun;88(6):1361-72. doi: 10.2106/JBJS.D.03018. PMID 16757774
- [Background] Sauerland S, Nagelschmidt M, Mallmann P, Neugebauer EA. Risks and benefits of preoperative high dose methylprednisolone in surgical patients: a systematic review. Drug Saf. 2000 Nov;23(5):449-61. doi: 10.2165/00002018-200023050-00007. PMID 11085349
- [Background] Holte K, Kehlet H. Perioperative single-dose glucocorticoid administration: pathophysiologic effects and clinical implications. J Am Coll Surg. 2002 Nov;195(5):694-712. doi: 10.1016/s1072-7515(02)01491-6. No abstract available. PMID 12437261
- [Background] Smeulers NJ, Wierda JM, van den Broek L, Gallandat Huet RC, Hennis PJ. Effects of hypothermic cardiopulmonary bypass on the pharmacodynamics and pharmacokinetics of rocuronium. J Cardiothorac Vasc Anesth. 1995 Dec;9(6):700-5. doi: 10.1016/s1053-0770(05)80232-0. PMID 8664462
- [Background] Hans P, Vanthuyne A, Dewandre PY, Brichant JF, Bonhomme V. Blood glucose concentration profile after 10 mg dexamethasone in non-diabetic and type 2 diabetic patients undergoing abdominal surgery. Br J Anaesth. 2006 Aug;97(2):164-70. doi: 10.1093/bja/ael111. Epub 2006 May 12. PMID 16698859
- [Background] Abdelmalak BB, Bonilla AM, Yang D, Chowdary HT, Gottlieb A, Lyden SP, Sessler DI. The hyperglycemic response to major noncardiac surgery and the added effect of steroid administration in patients with and without diabetes. Anesth Analg. 2013 May;116(5):1116-1122. doi: 10.1213/ANE.0b013e318288416d. Epub 2013 Apr 4. PMID 23558840
- [Background] Bailey IS, Karran SE, Toyn K, Brough P, Ranaboldo C, Karran SJ. Community surveillance of complications after hernia surgery. BMJ. 1992 Feb 22;304(6825):469-71. doi: 10.1136/bmj.304.6825.469. PMID 1547415
- [Background] Maldonado CC, Bentley AJ, Mitchell D. A pictorial sleepiness scale based on cartoon faces. Sleep. 2004 May 1;27(3):541-8. doi: 10.1093/sleep/27.3.541. PMID 15164912